CLINICAL TRIAL: NCT05721625
Title: Comparison of the Effects of Aerobic Exercise and Connective Tissue Massage in Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/02/01
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Women
Keywords: sleep, depression, massage, exercise
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The aerobic exercise program will be applied at moderate intensity 3 days a week for 8 weeks. Walking will be recommended as an aerobic exercise
  Interventions: Other: Aerobic exercise
- Massage group (Active Comparator): Connective tissue massage will be applied by the physiotherapist 3 days a week for 8 weeks. While postpartum women are in the sitting position, this massage will be applied on whole back.
  Interventions: Other: Connective tissue massage

INTERVENTIONS:
Other: Aerobic exercise — The aerobic exercise program will be applied at moderate intensity 3 days a week for 8 weeks. Walking will be recommended as an aerobic exercise
  Arms: Exercise group
Other: Connective tissue massage — Connective tissue massage will be applied by the physiotherapist 3 days a week for 8 weeks. While the patients are in the sitting position, this massage will be applied on whole back.
  Arms: Massage group

SUMMARY:
The aim of this study is to compare the effects of aerobic exercise and connective tissue massage on sleep, mother-infant attachment and psychological state in postpartum women.

DETAILED DESCRIPTION:
Postpartum period can affect the mental and physical health of women. Women may experience sleep problems and psychological problems due to hormonal changes and newborn care responsibilities. As a result, mother-infant attachment may also be affected. Physical activity and exercise should be encouraged in the postpartum period. It is known that aerobic exercises have positive effects on sleep and psychological problems. With the effects of connective tissue massage on the autonomic and circulatory system in the body, positive effects on sleep and psychological state can be achieved, but there are insufficient studies on this subject. In addition, no study has been found to the best of our knowledge comparing the effects of aerobic exercise and connective tissue massage in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum 6th week-1 year
* Between the ages of 18-45
* Being literate

Exclusion Criteria:

* Those with orthopedic, neurological, rheumatological, mental or any systemic chronic diseases
* Those with cardiac problems that may interfere with exercise
* Those with suspected pregnancy
* Those with malignancy
* Those who have infection
* Those who do not regularly participate in the treatment program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 40 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Postpartum Sleep Quality Scale | change from baseline at 8 weeks
  In order to measure Postpartum Sleep Quality, Postpartum Sleep Quality Scale will be used. The scale includes 14 items. The lowest score that can be obtained from the scale is 0, and the highest score is 56. An increase in the score indicates a decrease in sleep quality.

SECONDARY OUTCOMES:
Mother to Infant Bonding Scale | change from baseline at 8 weeks
  The Mother to Infant Bonding Scale, which was developed to be applied to the mother from the first day immediately after birth and allows the mother to express her feelings towards her baby in one word, will be used. This scale consists of 8 items. The lowest score that can be obtained from the scale is 0 and the highest score is 24. As the score obtained from the scale increases, the level of mother-infant attachment decreases.
Edinburgh Postpartum Depression Scale | change from baseline at 8 weeks
  The Edinburgh Postpartum Depression Scale, which was prepared for screening purposes to determine the risk of depression in postpartum women, is not intended to diagnose depression. This scale consists of 10 items. The lowest score that can be obtained from the scale is 0 and the highest score is 30. The cut-off point of the scale was calculated as 13, and women with a scale score of 13 or more were considered as the risk group.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Study Director — Ankara Yildirim Beyazıt University